CLINICAL TRIAL: NCT05998317
Title: Dexamethasone At-induction vs At-night to Prevent Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy: A Protocol for Randomized Clinical Trial
Brief Title: Dexamethasone at Night vs at Induction on PONV After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R.23.07.2239
Record Dates: First submitted 2023-08-11; First posted 2023-08-18 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Nausea and Vomiting; Postoperative Pain; Laparoscopic Cholecystectomy
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial superiority parallel trial. This is a pilot trial and the sample size will be updated after the pilot study completion and the approval of the local Institutional Review Board (IRB).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The pharmacists will prepare the study drug, either dexamethasone or saline in 10 mL similar syringes, according to the allocation. The syringe will be labeled with the patient's name and the allocation group, A or B. The study participants, caregivers, data collectors, and data analysts will all be blinded. The pharmacists will not participate in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- At-night dexamethasone (Experimental): Patients in the intervention group will receive intravenous 8 mg dexamethasone at night before surgery. The time of dexamethasone administration will be recorded. The dexamethasone ampule will be diluted in a 10 ml syringe and given in at least one minute to avoid unpleasant sensation in injection.
  Interventions: Drug: At-night Dexamethasone
- At-induction dexamethasone (Active Comparator): Patients in the control group will receive intravenous 8 mg dexamethasone just before or at the induction of anesthesia. The dexamethasone ampule will be diluted in a 10 ml syringe and given in at least one minute to avoid unpleasant sensation in injection.
  Interventions: Drug: At-induction Dexamethasone

INTERVENTIONS:
Drug: At-night Dexamethasone — Patients in the intervention group will receive intravenous 8 mg dexamethasone at night before surgery. The time of dexamethasone administration will be recorded. The dexamethasone ampule will be diluted in a 10 ml syringe and given in at least one minute to avoid unpleasant sensation in injection.
  Arms: At-night dexamethasone
Drug: At-induction Dexamethasone — Patients in the control group will receive intravenous 8 mg dexamethasone just before or at the induction of anesthesia. The dexamethasone ampule will be diluted in a 10 ml syringe and given in at least one minute to avoid unpleasant sensation in injection.
  Arms: At-induction dexamethasone

SUMMARY:
Since the peak effect of the dexamethasone is delayed to 12-16 hours after iv administration, we designed this study to investigate the effect of administering dexamethasone at-night before surgery versus at-induction (the standard timing) in prevention of postoperative nausea and vomiting after laparoscopic cholecystectomy.

A pilot randomized controlled study (60 cases) will be started to explore the potential difference, ensure correct and rigorous data collection, and calculate the sample size for a larger pragmatic trial.

DETAILED DESCRIPTION:
Background:

Postoperative nausea and vomiting (PONV) are common complications after laparoscopic cholecystectomy. The aim of this study is to evaluate the efficacy of administration of prophylactic dexamethasone 12-hours prior to induction of anesthesia in preventing PONV after elective laparoscopic cholecystectomy, as it reaches its peak effect at 2-12 hours and lasts for 72 hours after intravenous (iv) administration.

Methods:

This is a parallel two-arm, randomized (1:1), double-blind, controlled, single-center trial. Adults (≥18 years) with American Society of Anesthesiology (ASA) physical status I-III scheduled for elective laparoscopic cholecystectomy will be eligible for inclusion. The participants will be randomized to receive either 8 mg IV Dexamethasone at time of induction of anesthesia or 8 mg IV Dexamethasone at 12 hours prior to induction of anesthesia. The primary outcome will be the incidence of postoperative nausea and vomiting. A total of 60 patients will be recruited as a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive adults (older than 18 years) with ASA physical status I-III undergoing elective laparoscopic cholecystectomy surgery at gastrointestinal surgery center.

Exclusion Criteria:

* patient refusal
* use of steroids or antiemetic agents within 1 week of surgery
* chronic opioid therapy
* history of allergy to any study medications
* serum creatinine > 1.4 mg/dl
* liver enzymes more than triple normal limits
* pregnancy
* psychiatric or neurologic diseases or socioeconomic status that would hinder postoperative quality of recovery questionnaire
* Patients whose laparoscopic surgery is converted to open surgery after enrollment will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-08 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
postoperative nausea or vomiting (PONV) | 24 hours after surgery
  incidence of PONV (binary outcome as yes/No)

SECONDARY OUTCOMES:
The need for rescue antiemetic | 24 hours after surgery
  Dichotomous yes/no outcome
The need for rescue analgesia | 24 hours after surgery
  Dichotomous yes/no outcome
Postoperative Care Unit (PACU) and Early PONV | within 6 hours after surgery
  Dichotomous yes/no outcome
Late PONV | 6-24 hours after surgery
  Dichotomous yes/no outcome
Visual Analogue Scale (VAS) | at the time of discharge from PACU (usually at 2 hours after surgery)
  VAS as a scale 0 - 10
Visual Analogue Scale (VAS) | at the time of discharge from hospital (usually 24 hours after surgery)
  VAS as a scale 0 - 10
Postoperative quality of recovery (QoR) | 24 hours after surgery
  QoR-15 questionnaire (doi: https://doi.org/10.1097/ALN.0b013e318289b84b)
Post-Discharge Nausea and Vomiting (PDNV) | at 72 hours after surgery
  evaluated by telephone by Dichotomous yes/no outcome

OTHER OUTCOMES:
Surgical Site Infection | at follow-up (usually at 7 days after surgery)
  infection as defined by the surgeon) at the trocar's or the drainage tube sites.
Itching or burning sensation | during injection of the dexamethasone
  as described by the patient as dichotomous outcome yes/no outcome

CONTACTS AND LOCATIONS:
Overall Officials: Moataz M Emara, MD, EDAIC, Study Chair — Mansoura University Faculty of Medicine
Locations (1):
- Faculty of Medicine, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The anonymised data will be available on appropriate response with the prinicipal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within one year of study completion
Access Criteria: will be notified shortly